CLINICAL TRIAL: NCT01134575
Title: Treatment of Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL) With CMC-544 (Inotuzumab Ozogamycin), With or Without Later Addition of Rituximab
Brief Title: CMC-544 in Relapsed Refractory Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0872; NCI-2011-01699 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2019-05-22 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Relapsed; Refractory; Acute Lymphoblastic Leukemia; ALL; Burkitt's lymphoma; Lymphoblastic lymphoma; CMC-544; Inotuzumab Ozogamycin; Rituxan; Rituximab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin; Rituximab

STUDY DESIGN:
Intervention Model Description: The study started as a single arm study of Inotuzumab Ozogamicin administered at two different dose levels. The protocol was later amended to modify to weekly Inotuxumab Ozogamicin administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 (Experimental): First patients > 16 years and < 16 years receive CMC-544 (Inotuzumab Ozogamycin) at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle. With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
  Interventions: Drug: CMC-544 (Inotuzumab Ozogamycin); Drug: Rituximab
- Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin) (Experimental): CMC-544 (Inotuzumab Ozogamycin) 0.8 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 1, 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 8, and 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 15. Weekly doses can be given at + 1 day. Course may be repeated every 3 weeks. Rituximab will be given on Day 1 and CMC-544 on Day 2 of the first dose; with subsequent weekly doses, both will be given weekly, rituximab preceding CMC-544. The weekly dose of rituximab will be 375 mg/m2.
  Interventions: Drug: CMC-544 (Inotuzumab Ozogamycin); Drug: Rituximab
- Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 (Experimental): First patients > 16 years and < 16 years receive CMC-544 (Inotuzumab Ozogamycin) at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle. With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
  Interventions: Drug: CMC-544 (Inotuzumab Ozogamycin); Drug: Rituximab

INTERVENTIONS:
Drug: CMC-544 (Inotuzumab Ozogamycin) — First patients > 16 years and < 16 years receive CMC-544 at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle.
  Part 2 CMC-544 (Inotuzumab Ozogamycin) 0.8 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 1, 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 8, and 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 15. Weekly doses can be given at + 1 day. Course may be repeated every 3 weeks. Rituximab will be given on Day 1 and CMC-544 on Day 2 of the first dose; with subsequent weekly doses, both will be given weekly, rituximab preceding CMC-544. The weekly dose of rituximab will be 375 mg/m2.
Drug: Rituximab — With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
  Other Names: rituxan

SUMMARY:
The goal of this clinical research study is to learn if CMC-544 given alone, and possibly given in combination with rituximab, can help to control the disease in patients with ALL. The safety of the study drug(s) will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

CMC-544 is a monoclonal antibody (a substance that can locate and bind to cancer cells). It is designed to attach to C22, a molecule that is found on most cancer cells with ALL. This may cause the cancer cells to die.

Rituximab is a monoclonal antibody that is designed to attach to leukemia cells and activate a series of events that may cause the cancer cells to die.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive CMC-544 by vein over about 60 minutes on Day 1 of each study "cycle" or over 60 minutes at a lowered dose on Days 1, 8 and 15 of each cycle, depending on when you joined the study. No matter what dosing schedule you are on, you will receive the same total dosage of CMC-544. Each study cycle is about 3-4 weeks.

If the disease is not responding to the CMC-544 after 2 cycles, you will begin receiving rituximab. On Day 1 of Cycle 3, you will receive rituximab by vein over about 8 hours. On Day 2 of Cycle 3, you will receive CMC-544 alone by vein over about 60 minutes. Then, starting on Day 1 of Cycle 4, you will begin receiving rituximab by vein over about 8 hours and CMC-544 by vein over about 60 minutes at least 2-4 hours after you receive the rituximab. You will receive this combination 1 time every week.

Your dose of the study drug(s) may change depending on any side effects you may have.

Study Visits:

You will have study visits within 1 week before Day 1 of each study cycle. At each study visit, the following tests and procedures will be performed:

* You will have a physical exam.
* Your performance status will be recorded.
* You will be asked how you are feeling and about any drugs you may be taking.
* You will have an ECG before you receive treatment with CMC-544 (+ 2 days).
* Blood (about 1 tablespoon) may be drawn to test how the study drug(s) may affect cancer cells before you receive the CMC-544 infusion.
* If you are receiving rituximab and if you have a history of irregular heartbeat or chest pain (due to heart trouble), you will have ECGs performed before the start of the rituximab, once during the infusion, and within 2 hours after the infusion. Rituximab infusion will be stopped if you experience any serious episodes of irregular heartbeat.
* If you are receiving rituximab, you may be examined for any signs or symptoms of bowel obstruction (blockage) and/or perforation (hole in the intestines, which may cause the contents to leak). Appropriate radiologic tests and surgical consults will be performed as needed.

Blood (about 1 tablespoon each time) will be drawn 1-3 times each week during Cycles 1 and 2, and at least 1 time every week during all other cycles for routine tests. Your doctor may decide to have more than 3 blood draws during Cycles 1 and 2.

You will have a bone marrow aspirate and/or biopsy between Days 14-21 (+/- 3 days) of Cycle 1 then every 1-2 cycles to check the status of the disease. You may have additional bone marrow aspirates and/or biopsies if your doctor feels it is necessary.

Length of Study:

You may receive CMC 544 with or without rituximab for up to 12 months. You will be taken off study if the disease gets worse or if you have intolerable side effects

Follow-up Visits:

You will have a follow-up visit 30 days after your last dose of the study drug(s). At this visit, you will be asked about any side effects you may be having. If you cannot make it to the clinic for this visit, it can be done over the phone with a member of the study staff. The phone call should last about 10 minutes.

This is an investigational study. Rituximab is FDA approved and commercially available for the treatment of lymphoid cancer. Neither CMC-544 nor the CMC-544/rituximab combination are FDA approved or commercially available. Their use in this study is investigational.

Up to 90 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Previously treated ALL (including Burkitt's lymphoma and lymphoblastic lymphoma) in relapse or primary refractory. Patients in first relapse will be eligible regardless of the first remission duration. At least 10 patients in Salvage 1-2 will be treated to assess anti-ALL response more precisely.
2. Age 16 years or older. Pediatric patients (<16 years old) will be allowed into the study after safety is established, that is at least 10 adult patients having received 1 or more cycles each.
3. Zubrod performance status 0-3.
4. Adequate liver function (bilirubin </= 1.5 mg/dL and Alanine transaminase (SGPT) or Aspartate transaminase (SGOT) </= 3 x upper limit of normal [ULN], unless considered due to tumor), and renal function (creatinine </= 2 mg/dL). Even if organ function abnormalities are considered due to tumor, the upper limit for bilirubin is </= 2.0 mg/dL and creatinine </= 3 mg/dL.
5. Male and female patients who are of childbearing potential agree to use an effective barrier method of birth control (e.g., latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 14 days of study start (applies only if patient is of childbearing potential. Non-childbearing is defined as >/= 1 year postmenopausal or surgically sterilized).

Exclusion Criteria:

1. Patient with active heart disease (NYHA class >/= 3 as assessed by history and physical examination).
2. Patients with a cardiac ejection fraction (as measured by either Radionuclide angiography (MUGA) or echocardiogram) < 45% are excluded.
3. Patients who receive other chemotherapy. Patients must have been off previous therapy for >/= 2 weeks and must have recovered from acute toxicity (to grade 1 or less) of all previous therapy prior to enrollment (consent signing). (Concurrent therapy for central nervous system [CNS] prophylaxis or treatment for CNS relapse is permitted). Treatment may start earlier if necessitated by the patient's medical condition (e.g. rapidly progressive disease) following discussion with the Principal Investigator.
4. Prior allogeneic stem cell transplant in previous 4 months.
5. Peripheral lymphoblasts > 50 x 10^9/L.
6. Pregnant and breast-feeding patients are excluded.
7. Patients with known hepatitis B are excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06-04 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Zhao Y, Short NJ, Kantarjian HM, Chang TC, Ghate PS, Qu C, Macaron W, Jain N, Thakral B, Phillips AH, Khoury J, Garcia-Manero G, Zhang W, Fan Y, Yang H, Garris RS, Nasr LF, Kriwacki RW, Roberts KG, Konopleva M, Jabbour EJ, Mullighan CG. Genomic determinants of response and resistance to inotuzumab ozogamicin in B-cell ALL. Blood. 2024 Jul 4;144(1):61-73. doi: 10.1182/blood.2024023930. PMID 38551807
- [Derived] Kantarjian H, Thomas D, Jorgensen J, Jabbour E, Kebriaei P, Rytting M, York S, Ravandi F, Kwari M, Faderl S, Rios MB, Cortes J, Fayad L, Tarnai R, Wang SA, Champlin R, Advani A, O'Brien S. Inotuzumab ozogamicin, an anti-CD22-calecheamicin conjugate, for refractory and relapsed acute lymphocytic leukaemia: a phase 2 study. Lancet Oncol. 2012 Apr;13(4):403-11. doi: 10.1016/S1470-2045(11)70386-2. Epub 2012 Feb 21. PMID 22357140
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: June 2010 to October 2012
Groups:
- Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2; Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2: First patients > 16 years and < 16 years receive CMC-544 (Inotuzumab Ozogamycin) at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle. With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
  CMC-544 (Inotuzumab Ozogamycin): First patients > 16 years and < 16 years receive CMC-544 at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle.
  Rituximab: With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
- Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin): CMC-544 (Inotuzumab Ozogamycin) 0.8 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 1, 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 8, and 0.5 mg/m^2 IV over 1 hour (+ 15 minutes) on Day 15. Weekly doses can be given at + 1 day. Course may be repeated every 3 weeks. Rituximab will be given on Day 1 and CMC-544 on Day 2 of the first dose; with subsequent weekly doses, both will be given weekly, rituximab preceding CMC-544. The weekly dose of rituximab will be 375 mg/m2.
  CMC-544 (Inotuzumab Ozogamycin): First patients > 16 years and < 16 years receive CMC-544 at a dose of 1.3 mg/m^2 by vein (IV) over 1 hour during Course 1, and 1.8 mg/m^2 IV over 1 hour during Course 2 and subsequently. In all other patients beginning dose of 1.8 mg/m^2 IV over 1 hour every 4 week cycle.
  Rituximab: With no improvement after 2 courses of CMC-544, addition of Rituximab dose 375 mg/m^2 IV (by vein) over 2-6 hours every 3-4 weeks.
Period: Overall Study
Arm/Group | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin)
Started | 3 | 45 | 42
Completed | 3 | 45 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin) | Total
Number analyzed (Participants) | 3 | 45 | 42 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 2 | 5
  Between 18 and 65 years | 2 | 33 | 30 | 65
  >=65 years | 1 | 9 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 32 [24 to 67] | 38 [6 to 80] | 51 [4 to 83] | 40 [4 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 24 | 15 | 39
  Male | 3 | 21 | 27 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5
  White | 3 | 33 | 35 | 71
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 3 | 45 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Response
Description: Primary endpoint for efficacy is response which is defined as: Complete Remission (CR), Complete Remission without recovery of counts (CRi) or Partial Remission (PR). Complete remission (CR): Disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x109/L, platelet count >100x109/L, and normal marrow differential (< 5% blasts). 8.2 Complete remission without recovery of counts (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 109/L; neutrophils < 1 x 109/L). Partial remission (PR): Peripheral blood count recovery as for CR, but with decrease in marrow blasts of > 50% and not more than 25% abnormal cells in the marrow.
Time Frame: After cycle 2, for up to 8 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin)
Number analyzed (Participants) | 3 | 45 | 42
Participants | 3 | 25 | 24

ADVERSE EVENTS:
Time Frame: Up to two years
Arm/Group | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin)
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/45 | 5/42
Serious Adverse Events (participants affected / at risk) | 2/3 | 26/45 | 10/42
Other Adverse Events (participants affected / at risk) | 3/3 | 29/45 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 (N=3) | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 (N=45) | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin) (N=42)
Abdominal Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Allergic Reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Bilateral Extremity Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bone Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to Thrive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 2 (2) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage CNS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Laparoscopic Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Leukemic CNS Involvement (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Neutropenic Fever (Infections and infestations) | 2 (2) | 15 (18) | 6 (9)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 6 (6) | 4 (5)
Bactremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: CMC-544 (Inotuzumab Ozogamycin) 1.3mg/m^2 (N=3) | Period 2: CMC-544 (Inotuzumab Ozogamycin) 1.8mg/m^2 (N=45) | Period 3: Weekly CMC-544 (Inotuzumab Ozogamycin) (N=42)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Abdominal Pain (General disorders) | 1 (1) | 9 (9) | 6 (6)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 5 (5) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back Pain (General disorders) | 0 (0) | 11 (12) | 2 (2)
Increased Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 5 (9) | 3 (3)
Blood Glucose Increased (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 6 (6) | 1 (1)
Chills (General disorders) | 1 (1) | 10 (12) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 6 (7) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 1 (1)
Creatinine Increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (4)
Dehydration (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (6) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 9 (10) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 4 (5) | 1 (1)
Dry Eye Syndrome (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 9 (10) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 9 (14) | 6 (6)
Fatigue (General disorders) | 1 (1) | 4 (7) | 2 (2)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 10 (16) | 3 (3)
Fecal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 15 (22) | 1 (1)
Gastrointestianl Other (Gastrointestinal disorders) | 0 (0) | 4 (5) | 2 (2)
Headache (General disorders) | 0 (0) | 15 (18) | 4 (4)
Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Hematoma (Blood and lymphatic system disorders) | 1 (3) | 2 (2) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 5 (5)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Hepatobiliary/Pancreas Other (Hepatobiliary disorders) | 0 (0) | 0 (0) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 4 (4) | 2 (2)
Hypotension (Cardiac disorders) | 0 (0) | 7 (8) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 4 (7) | 3 (3)
Insomnia (General disorders) | 0 (0) | 1 (1) | 3 (3)
Intracranial Hemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Localized Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Lymphatics Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Lymphedema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Metabolic/Laboratory (Metabolism and nutrition disorders) | 0 (0) | 8 (16) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 10 (13) | 7 (8)
Neck Pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Neurology (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0)
Ocular/Visual Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Oral Hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Pain (General disorders) | 1 (1) | 11 (20) | 2 (2)
Pain Extremity (General disorders) | 1 (1) | 12 (14) | 4 (4)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 3 (4)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 4 (4)
Pneumonia (Infections and infestations) | 0 (0) | 6 (6) | 9 (9)
Pneumonitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Other (Reproductive system and breast disorders) | 1 (1) | 6 (8) | 3 (3)
Rash Desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Rectal Pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Renal/Genitourinary Other (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 3 (4) | 1 (1)
Serum Calcium Decreased (Metabolism and nutrition disorders) | 0 (0) | 8 (8) | 0 (0)
Serum Glucose Decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Serum Magnesium Decreased (Metabolism and nutrition disorders) | 0 (0) | 9 (11) | 0 (0)
Serum Phosphate Decreased (Metabolism and nutrition disorders) | 1 (2) | 8 (12) | 0 (0)
Serum Potassium Increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Serum Sodium Decreased (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 0 (0)
Serum Potassium Decreased (Metabolism and nutrition disorders) | 0 (0) | 12 (17) | 2 (2)
Sinus Bradycarida (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 5 (5) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Toothache (General disorders) | 0 (0) | 1 (1) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (11) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-12-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT01134575/Prot_SAP_000.pdf